CLINICAL TRIAL: NCT05561634
Title: Evaluation of Radiotherapy After Complete Response to Sonic Hedgehog Pathway Inhibitors in Patients With Locally Advanced Basal Cell Carcinoma: a Prospective Multicenter Study
Brief Title: Radiotherapy by Sonic Hedgehog Pathway Inhibitors in Basal Cell Carcinoma
Acronym: RADIOSONIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021_0710; 2022-A01424-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Basal Cell Carcinoma; Radiotherapy; Complications
Keywords: Locally advanced basal cell carcinoma; Sonic Hedgehog inhibitors; Consideration radiotherapy
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Radiotherapy; Observation; HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHHI then follow-up (Sham Comparator)
  Interventions: Radiation: Radiotherapy; Other: Observation
- SHHI then radiotherapy (Experimental)
  Interventions: Radiation: Radiotherapy; Drug: Vismodegib

INTERVENTIONS:
Radiation: Radiotherapy — Irradiation of the tumoral bed.
Other: Observation — Patients will be followed up in consultation every 3 months.
  Arms: SHHI then follow-up
Drug: Vismodegib — Sonic Hedgehog inhibitors (SHHi) = Vismodegib et Sonidegib,
  Arms: SHHI then radiotherapy

SUMMARY:
Locally advanced basal cell carcinoma (BCC) are large BCCs or BCCs located in areas subject to functional and aesthetic risk following surgery or radiotherapy. In these particular situations, surgery and radiotherapy are sometimes not appropriate, and Sonic Hedgehog inhibitors (SHHi) (Vismodegib and Sonidegib) can be proposed. SHHi are effective treatments in laBCC but most CR patients discontinue treatment because of tolerability. Approximately 65% of the population experience a relapse after discontinuation. A few cases of patients treated concomitantly by radiotherapy and vismodegib have been reported in the literature, suggesting that combining vismodegib and concomitant radiotherapy results in an improved overall response compared to a single modality treatment. There is no study evaluating a "consolidation radiotherapy" after complete response to SHHi. We carry out a prospective multicenter study in order to evaluate consolidation radiotherapy in patients with laBCC after achieving complete response with SHHi, with the hypothesis of reducing recurrence after discontinuation of SHHi.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years
* Locally advanced non-recurrent BCC in complete response after first course of SHHi
* Complete response has to be confirmed histologically
* Available photography or CT scan before SHHi treatment allowing delineation of the initial tumor

Exclusion Criteria:

* Patients with distant metastasis
* Patients with Gorlin's syndrome
* Prior radiotherapy to the region of the studied cancer that would result in overlap of radiation therapy fields
* Pregnant women
* Life expectancy less than 1 year
* Inability to receive informed consent
* Inability to participate in the entire study
* Lack of social security coverage
* Refusal to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2029-06-20 (Estimated); Study Completion 2029-06-20 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a local relapse at 2 years in both groups. | At 2 years

SECONDARY OUTCOMES:
Occurrence of local relapse at 1 and 3 years. | at 1 year and at 3 years
Occurrence of adverse effects in the radiotherapy group. | at 1 year, at 2 years and at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Mortier, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU Lille, Lille, France